CLINICAL TRIAL: NCT02656888
Title: Phase III, National, Multicenter, Randomized, Double Blind Clinical Trial to Evaluate the Efficacy and Safety of Irlanda-1-Association on the Treatment of Common Cold in Children
Brief Title: Efficacy and Safety of Irlanda-1-Association on the Treatment of Common Cold in Children
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMS0615
Record Dates: First submitted 2016-01-12; First posted 2016-01-15 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Common Cold
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irlanda-1-Association (Experimental): For children 2 to 6 years old: take 2,5 mL every 12 hours (2x/day), oral route. For children 6 to 12 years old: take 5 mL every 12 hours (2x/day), oral route. For children 12 to 17 years old: take 10 mL every 12 hours (2x/day), oral route.
  Interventions: Drug: Irlanda-1-Association
- Placebo (Placebo Comparator): For children 2 to 6 years old: take 2,5 mL every 12 hours (2x/day), oral route. For children 6 to 12 years old: take 5 mL every 12 hours (2x/day), oral route. For children 12 to 17 years old: take 10 mL every 12 hours (2x/day), oral route.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Irlanda-1-Association — For children 2 to 6 years old: take 2,5 mL every 12 hours (2x/day), oral route. For children 6 to 12 years old: take 5 mL every 12 hours (2x/day), oral route. For children 12 to 17 years old: take 10 mL every 12 hours (2x/day), oral route.
  Other Names: EMS association
  Arms: Irlanda-1-Association
Drug: Placebo — For children 2 to 6 years old: take 2,5 mL every 12 hours (2x/day), oral route. For children 6 to 12 years old: take 5 mL every 12 hours (2x/day), oral route. For children 12 to 17 years old: take 10 mL every 12 hours (2x/day), oral route.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy of the drug associations in the treatment of common cold symptoms.

DETAILED DESCRIPTION:
Double-blind,randomized, multicenter; Maximal experiment duration: 7 days; 03 visits; Safety and efficacy evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Participant within 48 hours of the onset of common cold symptoms: headache, sneezing, sore throat, nasal obstruction, cough, coryza and body pain;
* Signed Consent of the patient;
* Participant whose tutors have the capacity to understand and consent to the child's participation in the clinical study, manifested by signing TCLE

Exclusion Criteria:

* Patients with any clinically significant disease that in the investigator is opinion can´t participate in the study;
* Patients with any laboratory finding or image finding that in the investigator is opinion can´t participate in the clinical trial;
* Patients with history of hypersensitivity to any of the formula compounds;
* Participation in clinical trial in the year prior to this study;
* Patients with vaccine reaction;
* Patients who have uncontrolled asthma however, participants in use of pulmonary corticosteroids (alone or in combination with other products) will be allowed if they are in stable dose and diagnosed with controlled asthma;
* Patients with gastroesophageal reflux, gastric or duodenal ulcer or other serious disease of the gastrointestinal tract;
* Patients with diabetes mellitus type I and II;
* Pregnancy or risk of pregnancy and lactating patients;
* Patients who were in use of drugs that can interfere with flu symptoms evaluation.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Determine the efficacy of Irlanda_1 association in the treatment of common cold symptoms. | 7 days

SECONDARY OUTCOMES:
Safety will be evaluated by the adverse events occurrences | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Allergisa, Campinas, São Paulo, Brazil